CLINICAL TRIAL: NCT03254719
Title: Care Outcomes for Chiropractic Outpatient Veterans Aim 3-pilot Trial
Brief Title: Care Outcomes for Chiropractic Outpatient Veterans
Acronym: COCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Collaborators: University of Iowa (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: COCOV-Aim #3; R34AT008427 (NIH)
Record Dates: First submitted 2017-07-24; First posted 2017-08-18 (Actual); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Low Back Pain; PTSD; Depression; Anxiety
Keywords: Low Back Pain; Chiropractic; Veterans; PTSD; Depression; Anxiety
MeSH Terms: conditions — Low Back Pain; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Chiropractic care will be administered by licensed DCs who are current employees of the Iowa City VA Health Care System (ICVAHCS). Participants will receive chiropractic care at a frequency of 1-2 visits per week for a duration up to 10 weeks, with the frequency and duration of care individualized within established VA parameters. For this trial, the minimum treatment dose is 1 visit to the DC, while the maximum treatment dose is 12 visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Other): All participants enrolled in the study will receive chiropractic care consistent with the usual chiropractic procedures for the management of chronic low back pain at the Iowa City VA Health Care System. Participants will also complete study assessments as described in outcomes.
  Interventions: Other: Study assessments

INTERVENTIONS:
Other: Study assessments — All participants will be asked to complete study assessments at baseline visit, and weeks 3, 5, 7, and 10. Study participants will receive spinal manipulation and appropriate adjunctive therapies provided by doctors of chiropractic.

SUMMARY:
The primary objectives of this pilot trial are to evaluate the feasibility, safety and acceptability of an integrative care pathway that includes chiropractic care, for the coordinated care for Veterans Administration (VA) patients with chronic low back pain (cLBP), with an emphasis on those with mental health comorbidity, in preparation for the conduct of an appropriately powered multi-site randomized controlled trial (RCT). The secondary objectives are to collect study outcomes at the baseline visit (BV) and at weeks 3, 5, 7, and 10 to: 1) assess the success of collecting outcomes; 2) determine the outcome measures to use in a future RCT; and 3) determine preliminary intervention effect sizes and variability to aid in sample size determination for a future RCT. The investigators hypothesize that chiropractic care offers relief for pain and mental health symptoms through the direct effects of treatment-focused CMT, as well as through the indirect, non-specific effects of the team-based relationship with the clinician.

This pilot study is a single-arm trial. All participants will be asked to complete study outcomes which include the Roland Morris Disability Questionnaire (RMDQ), LBP intensity and interference as measured by the Defense and Veterans Pain Rating Scale (DVPRS), as well as the Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder 7-item Scale (GAD-7), Alcohol Use Disorders Identification Test (AUDIT), Post-traumatic Stress Disorder Checklist-Civilian Version (PLC-C), self-care behaviors, Keele Start Back Screening Tool (STarT Back), Healing Encounters and Attitudes Lists (HEAL), Expectations for Complementary and Integrative Treatments Questionnaire (EXPECT), and Pain Intensity, Enjoyment of Life, General Activity Assessment Tool (PEG) questionnaires, and the Pain Assessment Screening Tool and Outcomes Registry (PASTOR) assessment, which includes measures of pain, disability, mental health, quality of life enjoyment and satisfaction. All participants will receive up to 10 weeks of chiropractic care and will complete outcome assessments at weeks 3, 5, 7, and 10 of the study.

DETAILED DESCRIPTION:
The coinciding problems of chronic pain and mental illness are of great concern for patients seeking care within the Department of Veterans Affairs (VA) healthcare facilities. Of the 5.7 million veterans treated in VA facilities in 2012, more than half reported chronic pain syndromes, including chronic low back pain (cLBP). Veterans also experience many mental health comorbidities, such as depression, anxiety, post-traumatic stress disorder (PTSD), and substance abuse. Veterans in pain are often managed using prescription drugs, including opioids, psychotropic medications, and sleep agents. Non-pharmacological treatments for chronic pain, which also may provide relief of mental health symptoms, may be welcomed complementary therapies for veterans suffering from these conditions.

Patients with musculoskeletal (MSK) pain and pain at multiple locations often report depression, anxiety and other mental health symptoms. Chronic pain may perpetuate mental health comorbidity as these conditions share common pathophysiological pathways. Research has shown that the non-specific effects of empathetic doctor communication and therapeutic alliance improves clinical outcomes. The investigators hypothesize that chiropractic care offers relief for pain and mental health symptoms through the direct effects of treatment-focused chiropractic manipulative therapy (CMT), as well as through the indirect, non-specific effects of the team-based relationship with the clinician.

However, chiropractic care is not delivered in isolation from other treatments within the VA. Thus, the investigators will test a feasible, effective, patient-centered, guideline-based, integrative care model that integrates chiropractic into VA Patient Aligned Care Teams (PACTs). This integrative care pathway will involve primary care providers, mental health professionals, and doctors of chiropractic (DCs) engaged in the treatment of veterans with cLBP, with or without mental health comorbidity. While DCs are providing services within VA in increasing numbers over the past 13 years, as with any new service, adoption and appropriate placement faces challenges. Many VA providers may know little about the clinical approaches used by DCs. Similarly, DCs may not be fully aware of the processes involved in the delivery of primary care services within VA or the healthcare needs of veterans with mental illness. The purpose of this pilot clinical trial is to evaluate the feasibility, safety and patient perceptions of an integrative care pathway, developed through a consensus-based process, for the coordinated care for VA patients with cLBP and mental health comorbidity.

As this is a pragmatic trial, chiropractic care will consist of usual chiropractic procedures for the management chronic low back pain (cLBP). Treatment approaches will be based on clinical evaluation, which may include diagnostic testing, to determine a working diagnosis, rule out pathology, and/or to screen for conditions requiring referral or other co-management. The investigators anticipate that chiropractic care often will include some form of chiropractic manipulative therapy (CMT). DCs will likely also recommend rehabilitative exercise, stretching, or nutritional and lifestyle advice based upon clinical findings and patient goals/preferences. The investigators will evaluate treatments through electronic health records (EHR) data abstraction following completion of chiropractic care at Week 10. As per typical VA care, DCs will monitor the participant's health status throughout the trial and initiate referrals as clinically indicated. Referrals to primary care and mental health providers will be consistent with the chiropractic integrated care pathway developed during a prior phase of the study. The investigators anticipate the most common communication and referral methods will occur through note-review and countersign procedures, which are already established among VA providers using the VA electronic health record, but may also occur in person or via phone conversations. Chiropractic care will be administered by licensed DCs who are current employees of the Iowa City VA Health Care System (ICVAHCS).

ELIGIBILITY:
Inclusion Criteria:

* Veterans age 18 years or older
* Self-reported chronic LBP
* Ability to sign informed consent form

Exclusion Criteria:

* Use of chiropractic care within the past 90 days
* Impaired cognitive ability
* Not a candidate for chiropractic care
* Not able to attend chiropractic appointments
* Identified as at risk for suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Goertz, DC, PhD, Principal Investigator — The Spine Institute for Quality; Cynthia Long, PhD, Principal Investigator — Palmer Center for Chiropractic Research (PCCR)
Locations (4):
- United States (4):
  - VA Community Based Outpatient Clinic, Coralville, Iowa
  - Palmer Center for Chiropractic Research, Davenport, Iowa
  - Iowa City Veterans Affairs Health Care System, Iowa City, Iowa
  - The Spine Institute for Quality, Oskaloosa, Iowa

IPD SHARING:
Plan to Share IPD: No
Feasibility/pilot study

REFERENCES:
- [Result] Lisi AJ, Salsbury SA, Hawk C, Vining RD, Wallace RB, Branson R, Long CR, Burgo-Black AL, Goertz CM. Chiropractic Integrated Care Pathway for Low Back Pain in Veterans: Results of a Delphi Consensus Process. J Manipulative Physiol Ther. 2018 Feb;41(2):137-148. doi: 10.1016/j.jmpt.2017.10.001. PMID 29482827
- [Derived] Long CR, Salsbury SA, Vining RD, Lisi AJ, Corber L, Twist E, Abrams T, Wallace RB, Goertz CM. Care Outcomes for Chiropractic Outpatient Veterans (COCOV): a single-arm, pragmatic, pilot trial of multimodal chiropractic care for U.S. veterans with chronic low back pain. Pilot Feasibility Stud. 2022 Mar 7;8(1):54. doi: 10.1186/s40814-022-01008-0. PMID 35256010
- [Derived] Salsbury SA, Twist E, Wallace RB, Vining RD, Goertz CM, Long CR. Care Outcomes for Chiropractic Outpatient Veterans (COCOV): a qualitative study with veteran stakeholders from a pilot trial of multimodal chiropractic care. Pilot Feasibility Stud. 2022 Jan 14;8(1):6. doi: 10.1186/s40814-021-00962-5. PMID 35031072

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Unknown | 1
  Race: White | 36
  Race: Multi-racial | 1
  Race: Declined to Answer | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 2
  Ethnicity: Not Hispanic or Latino | 38
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Duration of Study Recruitment
Description: As part of the feasibility assessment, the investigators will monitor the amount of time it takes to complete study recruitment and enrollment, and data collection. The investigators will monitor this through a data capture program.
Time Frame: From date of first participant enrolled to date last participant is enrolled, up to 8 months.
Measure: Number; unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
months | 6

2. Primary Outcome: Diversity of Patient Demographics
Description: As part of the recruitment plan, investigators are trying to target female and minority veterans. Historically these groups have been underrepresented in veteran research. The investigators will review EHR data for participant demographics.
Time Frame: Screening through baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
Participants
  Multi-racial | 1
  White | 36
  Other or unspecified | 3
  Hispanic or Latino | 2
  Male | 31
  18-35 years | 6
  36-54 years | 16
  55+ years | 18

3. Primary Outcome: Number of Participants Engaged in Use of MyHealthEVet
Description: As part of the feasibility assessment, investigators will monitor the number of study participants who enroll in and have at least one communication with MyHealthEVet. MyHealthEVet is an online communication tool designed to partner veterans and the veteran's health care team. It provides information on the veteran's health record and health topics as well as allows messaging communication between veterans and health care providers. Usage reports generated by MyHealthEVet will be analyzed to determine number of study participants engaged.
Time Frame: 10 weeks from Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
Participants | 15

4. Primary Outcome: Acceptability
Description: Acceptability will be assessed by conducting structured, qualitative exit interviews with participants and providers.
Time Frame: At Week 10 of the study
Population: Acceptability of chiropractic service delivery as viewed by those veterans who were interviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 24
Participants
  Viewed as Positive | 10
  Viewed as Mixed Positive/Negative | 9
  Viewed as Negative | 5

5. Primary Outcome: Number of Participants With Reported Adverse Events
Description: Safety for this study will be assessed by the number of adverse events counted and recorded.
Time Frame: 10 weeks from Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
Participants | 6

6. Primary Outcome: Percentage of Participants Who Did Not Attend the Initial Chiropractic Visit, Withdrew, or Are Lost to Follow-up
Description: As part of the feasibility assessment and ability to calculate a sample size for a full scale trial with subgroup analysis, investigators will monitor the percentage of missing data. This will include the percentage of participants who did not attend the initial chiropractic visit and withdraw or are lost to follow-up.
Time Frame: 10 weeks from Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
Participants | 8

7. Secondary Outcome: Roland Morris Low Back Pain Disability Questionnaire (RMDQ)
Description: The RMDQ is a widely used health status measure for low back pain. Scoring of the RMDQ ranges from 0-24, with a higher score indicating an increase in low back pain disability. (0-24, 0=No Disability, 24=Severe Disability)
Time Frame: Baseline visit and weeks 5 and 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
score on a scale
  Baseline | 12.9 (5.1)
  Week 5 | 10.2 (5.5)
  Week 10 | 9.6 (6.2)

8. Secondary Outcome: Pain Assessment Screening Tool and Outcomes Registry (PASTOR)
Description: PASTOR is an on-line data collection tool based on the NIH Patient Reported Outcomes Measurement Information System (PROMIS) and adopted by the DoD/VA Pain Management Task Force. Specific measures include the Defense & Veterans Pain Rating Scale (DVPRS), an enhanced 11-item (total range 0-10, 0=no pain, 10=worst pain) numeric rating scale (NRS) that improves on standard pain NRS by including a Faces Rating Scale component; 'traffic light' color-coding system to delineate mild, moderate and severe pain; and word descriptors, paired with 4, 0-10 NRS items to quantify the impact of pain on general activity, sleep, mood, and stress. PASTOR incorporates PROMIS measures for mental health conditions (PTSD, depression, anxiety, anger, and alcohol use), physical and social function, fatigue, and pain interference with daily activities to provide graphical representation of improvements or declines in patient status that are compared to matched US samples on age, race/ethnicity and sex.
Time Frame: Baseline visit and weeks 5 and 10
Population: There are missing data when a participant was lost to follow-up or chose not to complete an item.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
score on a scale
  Worst Pain, Baseline | 6.4 (1.7)
  Worst Pain, Week 5: number analyzed (Participants) | 33
  Worst Pain, Week 5 | 5.7 (2.0)
  Worst Pain, Week 10: number analyzed (Participants) | 29
  Worst Pain, Week 10 | 5.3 (2.2)
  Average Pain, Baseline | 5.4 (1.4)
  Average Pain, Week 5: number analyzed (Participants) | 33
  Average Pain, Week 5 | 4.8 (1.8)
  Average Pain, Week 10: number analyzed (Participants) | 29
  Average Pain, Week 10 | 3.9 (2.0)

9. Secondary Outcome: STarT Back Screening Tool
Description: This is a 9-item, validated tool developed by Keele University to be used as a screening tool for patients with low back pain. It stratifies patients based on their prognosis of persistent disabling symptoms and allows practitioners to group patients into 3 categories (low, medium, or high risk of poor outcome).
Time Frame: Baseline visit and week 10
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
Participants
  Baseline: Low Risk | 2
  Baseline: Medium Risk | 17
  Baseline: High Risk | 13
  Baseline: Missing | 8
  Week 10: Low Risk | 9
  Week 10: Medium Risk | 12
  Week 10: High Risk | 7
  Week 10: Missing | 12

10. Secondary Outcome: Self-Efficacy for Managing Symptoms (SF8a)
Description: Developed by the Patient-Reported Outcomes Measurement Information System (PROMIS), this 8-item, self-reported tool will assess a person's level of confidence to manage/control symptoms, to manage their symptoms in different settings and to keep symptoms from interfering with work, sleep, relationships or recreational activities. Each question usually has five response options ranging in value from 1 to 5. The total raw score for a measure is converted to into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. A higher PROMIS T-score represents more of the concept being measured. For example, a T-score of 55 on the PROMIS Self-Efficacy for Managing Symptoms indicates that the respondent has greater self-efficacy for managing their symptoms than the general chronic condition population (half a standard deviation higher).
Time Frame: Baseline visit and week 10
Population: PROMIS - Self-Efficacy for Managing Symptoms - T score at Baseline and Week 10 follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 32
score on a scale
  Baseline | 41.6 (6.4)
  Week 10 | 43.5 (8.2)

11. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: This instrument is self-reported with nine items and will be used to assess depressive disorder. Total scores range from 0 to 27 with a score of 10-14 considered to be in the moderate range (0-27, 0=No Depression, 27=Severe Depression). It has been tested in primary care settings and has a test-retest reliability of 0.81 to 0.96.
Time Frame: Baseline visit and week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
score on a scale
  Baseline | 9.7 (5.6)
  Week 10 | 8.6 (5.8)

12. Secondary Outcome: Generalized Anxiety Disorder-7 (GAD-7)
Description: This instrument is self-reported with seven items and will be used to assess generalized anxiety disorder. At a cut off score of 10 (0-21, 0=No Anxiety Disorder, 21=Severe Anxiety Disorder), it has a sensitivity of 0.89 and specificity of 0.82 for identifying patients with GAD in primary care settings.
Time Frame: Baseline visit and week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
score on a scale
  Baseline | 7.7 (5.6)
  Week 10 | 6.8 (5.3)

13. Secondary Outcome: Alcohol Use Disorders Identification Test (AUDIT)
Description: Developed by the World Health Organization (WHO), this 10-item screening questionnaire determines harmful or hazardous consumption of alcohol, correctly classifying 95% of people as having a clinical diagnosis of an alcohol abuse disorder (0-12, 0=No Alcohol Use).
Time Frame: Baseline visit and week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
score on a scale
  Baseline | 2.2 (2.8)
  Week 10 | 1.7 (1.9)

14. Secondary Outcome: PTSD Checklist-Civilian (PCL-C)
Description: This 17-item, self-reported instrument will assess PTSD. A total severity score is determined by summing scores from each of 17 items. A change of 5-10 points represents the minimum threshold for determining treatment response; a 10-20 point change represents a clinically significant change in PTSD symptom severity (17-85, 17=Not at all Severe PTSD Symptoms, 85=Extremely Severe PTSD Symptoms).
Time Frame: Baseline visit and week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
score on a scale
  Baseline | 40.3 (18.1)
  Week 10 | 40.1 (19.3)

15. Secondary Outcome: Healing Encounters and Attitudes Lists (HEAL)
Description: HEAL is a validated item-bank comprised of 6 domains developed through the Patient Reported Outcomes Measurement Information System (PROMIS) methodology. Investigators will use HEAL to assess nonspecific factors known to influence patient outcomes, including perceptions of the patient-provider connection, healthcare environment, treatment expectancy, spirituality, positive or negative outlook, and attitudes toward complementary and alternative medicine (CAM). A higher T-score represents more of the concept being measured. A T-score of 50 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of more positive perception. For example, a T-score of 55 on Patient-Provider Connection indicates that the respondent has a more positive perception toward the patient-provider connection than the general chronic condition population (half a standard deviation higher).
Time Frame: After the initial chiropractic visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 29
score on a scale
  Patient-Provider Connection - T-Score | 60.9 (10.6)
  Healthcare Environment - T-Score | 54.4 (8.4)
  Treatment Expectancy - T-Score | 54.6 (11.5)
  Positive Outlook - T-Score | 52.0 (10.4)
  Spirituality - T-Score | 50.9 (13.3)
  Attitudes toward CAM - T-Score | 56.0 (9.6)

16. Secondary Outcome: Pain, Enjoyment, and General Activity (PEG)
Description: The PEG is a 3-item tool to improve assessment and monitoring of chronic pain. The overall PEG-3 score ranges from 0-10 with 10 indicating more pain, more interference with enjoyment of life, and more interference with general activity. Questions assess average pain intensity (P) (AVERAGE pain in past week: 0-10, 0= No Pain, 10=Pain as bad as you can imagine), interference with enjoyment of life (E), and interference with general activity (G) (In past week, how pain interfered with...(0-10, 0=Does not interfere, 10=Completely interferes).
Time Frame: Week 3 and Week 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 35
score on a scale
  Average pain, Week 3 | 5.1 (2.0)
  Average pain, Week 7 | 4.8 (2.0)
  Enjoyment of Life Pain Interference, Week 3 | 5.3 (2.2)
  Enjoyment of Life Pain Interference, Week 7 | 4.7 (2.5)
  General Activity Pain Interference, Week 3 | 5.2 (2.2)
  General Activity Pain Interference, Week 7 | 4.7 (2.7)
  Overall PEG-3 Score, Week 3 | 5.2 (2.0)
  Overall PEG-3 Score, Week 7 | 4.7 (2.3)

ADVERSE EVENTS:
Time Frame: Baseline to 10 weeks.
Description: An AE is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an IMP, regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 5/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=40)
Muscle pain (Musculoskeletal and connective tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT03254719/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT03254719/Prot_SAP_001.pdf